CLINICAL TRIAL: NCT03584022
Title: A Clinical Trial to Assess the Safety of a Novel Scaffold Biomaterial
Brief Title: Clinical Trial to Assess the Safety of a Novel Scaffold Biomaterial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anthony J. Windebank, Professor of Neurology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-008763
Record Dates: First submitted 2018-05-11; First posted 2018-07-12 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Neuropathy; Chronic Inflammatory Demyelinating Polyradiculoneuropathy; Vasculitic Neuropathy (Disorder); Amyloidosis; Hereditary Neuropathy; Sarcoid Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Amyloidosis | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: Patients planned for diagnostic sural nerve biopsy will be screened. Nerve conduction study of the sural nerve is part of standard of care for patients who are screened for the study. If the amplitude of sensory nerve action potential (SNAP) is equal to or greater than 2 μV and the patient meets the other inclusive criteria, the patient will be recruited to enter the study. Ultrasonography of the sural nerve will be conducted. If the diameter of the sural nerve is greater than 2.75mm, the patient will be assigned to the control group. If sural nerve diameter is equal to or smaller than 2.75mm, the patient will be randomized to either the control or study group. A study team member (clinical coordinator) will draw a number from an envelope that holds equal amount of odd and even numbers. If the number drawn is an odd number, the patient will be assigned to the control group. If the number drawn is an even number, the patient will be assigned to the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Biopsy + Nerve Repair (Experimental): Subjects will undergo standard sural nerve biopsy plus repair of the 6 cm nerve defect using a synthetic polymer (PCLF) nerve tube.
  Interventions: Device: Biopsy + Nerve Repair
- Biopsy Only (Sham Comparator): Subjects will undergo the same standard sural nerve biopsy procedure as the Experimental Group, but will not include the nerve repair.
  Interventions: Procedure: Biopsy Only

INTERVENTIONS:
Device: Biopsy + Nerve Repair — During the standard sural nerve biopsy procedure, a single-use, biodegradable implant designed to repair damaged peripheral nerves will be used to repair the nerve. The MCNS1 is a hollow nerve tube made of poly(caprolactone-fumarate) (PCLF), to connect severed nerve ends and promote the growth of regenerating axons.
  Arms: Biopsy + Nerve Repair
Procedure: Biopsy Only — Standard sural nerve biopsy only, without nerve repair.
  Arms: Biopsy Only

SUMMARY:
This is safety study. Subjects will be undergoing the surgical procedure of nerve biopsy. After routine surgery without grafting, patients develop swelling, redness, tenderness and dysesthesia at the biopsy site. In order to determine whether grafting is safe compared to not repairing the nerve, it is necessary to compare treated vs. untreated patients using systematic, sensitive and reproducible criteria.

DETAILED DESCRIPTION:
Patients will be evaluated for eligibility and then, after gaining informed consent, the surgical procedure will be scheduled. Baseline evaluations include physical/neurological examination, nerve conduction study and ultrasonography of the sural nerve, and testing for erythrocyte sedimentation rate, C-reactive protein and complete blood counts (with white blood cell differential). Surgery is done in an operating room under local or monitored anesthesia, depending on patient preference. An incision will be made above the ankle. Immediately after the surgery, the patient will repeat the baseline physical/neurological exams, and sural nerve ultrasonography.

Participants will be evaluated either in the clinic or by phone on a regular basis and will be required to keep a journal and fill out symptom questionnaires for up to 12 months post-procedure.

Development of a grade 4 local reaction at any time will fulfill criteria for review by the Data and Safety Monitoring Board (DSMB) for implant removal and definition as a failure.

ELIGIBILITY:
Inclusion Criteria

* Are between the ages of 18-75 years
* Have clinical indications for whole sural nerve biopsy
* Have a sural nerve SNAP with amplitude > or = 2 microvolt (μV)
* Are able to comply with protocol requirements
* Can provide written informed consent
* Willingness to complete study procedures

Exclusion Criteria

* Current smoker.
* History of prior musculoskeletal (joint or soft tissue) infection.
* Pre-operative nares culture positive for methicillin-resistant Staphylococcus Aureus (MRSA) or methicillin-sensitive Staphylococcus Aureus (MSSA)
* Have systemic immune disorders, such as Crohn's Disease, rheumatoid arthritis, or psoriasis with the exception of hyper/hypothyroidism.
* Have diabetes mellitus.
* Have previous trauma to the biopsy site.
* Have any major, clinically significant medical condition (e.g., within six months of baseline, had myocardial infarction, angina pectoris, and/or congestive heart failure) that, in the opinion of the investigator, would compromise the safety of patient.
* Are pregnant or breast-feeding.
* Unwilling to use adequate contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety as determined by number of participants with post-surgical reactions | up to 5 years post surgery
  Post-surgical reactions will include evaluations of the following:
  1. Percussion tenderness at site of proximal stump or repair site;
  2. Skin redness at the site of biopsy (length and width measured with calipers);
  3. Development of mild or moderate swelling along the site (yes or no). It is anticipated that this will resolve to a lower grade or progress to grade 4.
  4. Development of severe swelling or pustules or evidence of tube extrusion or wound dehiscence.

SECONDARY OUTCOMES:
Neuropathic pain as measured by SNAP | 3 months & 12 months
  Sensory nerve action potential (SNAP) will be measured at the ankle using small electric shocks and recording pads on the skin. This will be done by an experienced and board-certified electrophysiologist.
Neuropathic pain as measured by visual analogue pain scale | weekly, monthly for first 3 months, then 12 months and yearly for 4 years
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints of 'No pain' and 'Pain as bad as it could possibly be'. The subject is asked to mark his or her pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark defines the subject's pain.
Neuropathic pain as measured by visual analogue pain assessment questionnaire | weekly, monthly for first 3 months, then 12 months and yearly for 4 years
  Subjects will be asked to check all of the following that apply: 1) fever, 2) unexplained or new joint aches and pain, 3) increased skin redness at or near the site of the biopsy, 4) increased swelling at or near the site of the biopsy, 5) some degree of pain or discomfort at or near the site of the biopsy
Neuroma formation | 3 months & 12 months
  Non-invasive nerve ultrasound will be performed to determine neuroma formation
Sensory nerve regeneration as measured by SNAP | 3 months & 12 months
  The amplitude of sensory nerve action potential (SNAP) will be used to determine sensory nerve regeneration
Sensory nerve regeneration as measured by ultrasound | 3 months & 12 months
  Non-invasive nerve ultrasound will be performed to determine sensory nerve regeneration

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Windebank, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No